CLINICAL TRIAL: NCT00801112
Title: Developing Bioimpedance (BIA) as a Tool for Fluid Management in Peritoneal Dialysis Patients: A Validation Study
Brief Title: Bioimpedance as a Tool for Fluid Management in Peritoneal Dialysis (PD) Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital of North Staffordshire (Other)
Collaborators: St. James's Hospital, Ireland (Other); Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Professor Simon Davies, University Hospital of North Staffordshire
Other Study IDs: BIA-001MC
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2008-12-03 (Estimated); Status verified 2008-12

CONDITIONS: Fluid Status; Peritoneal Dialysis
Keywords: Bioimpedance; Fluid status; Peritoneal Dialysis; Extra-cellular fluid volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, urine and peritoneal fluid.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: PD patients with residual renal function >200ml with BIA monitor.
- 2: PD patients with residual renal function <200ml with BIA monitor.
- 3: PD patients with residual renal function >200ml without BIA monitor
- 4: PD patients with residual renal function <200ml without BIA monitor

SUMMARY:
Hypothesis: The investigators hypothesize that regular monitoring of BIA adds value to the management of fluid status in PD patients

Objectives of the study: The objective is to show that in patients where the additional information of body composition is available to the clinician that the ECFv is maintained within pre-agreed limits, ~ 1 liter, over the observation period of 12 months.

SCIENTIFIC BACKGROUND:

Low peritoneal ultrafiltration, and by inference low sodium removal, is associated with worse outcomes in PD. Equally, excessive fluid removal is a risk factor for dehydration and loss of residual renal function. Current guidelines have advocated a daily UF volume of 1litre; their blunt application could lead to either inappropriate early loss of residual function or modality transfer. There is a significant need for evidence on how to best manage fluid status in PD patients, both in terms of an appropriate clinical strategy and also a simple but reproducible tool to guide clinicians in how to apply this strategy.

It is likely that BIA will become the standard tool to aid clinicians in assessing fluid status. It is simple to perform, intervention studies have demonstrated its ability to identify changes in fluid status in response to changes in therapy and it is a powerful predictor of patient survival. There is, however a clear need at this stage for proof of principle studies to establish its true potential for added value in the routine management of patients.

Body composition changes spontaneously with time on PD. Short term changes in hydration (specifically extracellular fluid volume, ECFv) combined with medium term changes in muscle and fat make it difficult for the clinician to be sure if fluid status is stable. It is anticipated that regular BIA measurements will aid the clinician in managing this problem over and above monitoring of weight and fluid status. By randomizing patients into two groups who have regular BIA measurements, one of which the BIA data is available to the clinician it will be possible to see if these spontaneous changes in body composition can be accounted for.

ELIGIBILITY:
Inclusion Criteria:

* All PD patients who are clinically stable

Exclusion Criteria:

* Patients planning discontinuation of PD within 6 months.
* Patients who are unable to give consent.
* Patients who have peritonitis the last 30 days prior to study enrollment.
* Patients who are pregnant.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Incident and prevalent PD patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-01; Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Extra-cellular Fluid Volume (ECFv) determined from BIA to be maintained within pre-agreed limit of 1 liter. | 12 months

SECONDARY OUTCOMES:
Blood pressure control and residual urine volume. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Simon J Davies, MD FRCP, Principal Investigator — University Hospital of North Staffordshire
Locations (1):
- University Hospital of North Staffordshire, Stoke-on-Trent, Staffordshire, United Kingdom